CLINICAL TRIAL: NCT04360252
Title: Gracie Diet for Gastroesophageal Reflux Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00248899
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Gastroesophageal Reflux; GERD
Keywords: GERD; Diet; Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gracie Diet (Experimental): Patients will have a nutritional consultation and will follow the Gracie diet for a month.
  Interventions: Other: Gracie Diet

INTERVENTIONS:
Other: Gracie Diet — The patient is going to have an encounter with the nutritionist (either face to face or by phone call) and she will provide patient with the requisite nutritional information and will guide patient on how to properly adhere to the diet.
  The session is designed to: answer patient questions, educate patients so that patients understand the underlying nutritional concepts that the diet is based upon, support patients by empowering the patients to make healthy nutritional choices consistent with the diet, educate patients regarding the appropriate combinations of healthy foods, and help patients to develop menu samples based on the Gracie Diet when there is interest.

SUMMARY:
The goal of this clinical trial is to learn if dietary changes can help improve gastroesophageal reflux disease (GERD) symptoms. The main question[s] it aims to answer whether the Gracie Diet is an option to treat GERD symptoms in individuals wish to discontinue standard doses of PPI and / or H2 receptor antagonists.

Participants will be taken off PPI and be placed on the Gracie Diet for 8 weeks. Information about the participants reflux symptoms and GERD health related quality of life will be collected to assess the effect of the diet.

DETAILED DESCRIPTION:
GERD, is a common and chronic world-wide disease. Cardinal symptoms of this condition are heartburn-regurgitation, and sometimes with extra-intestinal symptoms that can affect patients' quality of life. Proton pump inhibitors (PPIs) potently inhibit gastric acid secretion and are widely used for treatment of acid-related diseases. This class of medications is the most widely used for the management of GERD. H2 Receptor Antagonists (H2RAs) are another type of medication used to of uncomplicated GERD, gastric or duodenal ulcers, gastric hypersecretion, and for mild to infrequent heartburn or indigestion. H2RAs decrease gastric acid secretion by reversibly binding to histamine H2 receptors located on gastric parietal cells, thereby inhibiting the binding and action of the endogenous ligand histamine.

Dietary modification is endorsed by the National Institutes of Health and the American College of Gastroenterology as a first-line therapy for patients with GERD. The Gracie Diet is thought to play an important role in the prevention of GERD. The concept behind this diet is that the consumption of proper food combinations promotes optimal health by preventing unhealthy chemical reactions in the digestive process such as fermentation and acidity.

This diet describes the benefits of combining different foods together and the downsides of combining others. It provides guidance on avoiding specific foods and combinations of foods that may aggravate GERD, and adopting meal spacing habits to improve overall health outcomes. The idea is that such dietary changes support more efficient digestion and encourage healthier lifestyles (i.e. smoking cessation, elimination of alcohol intake, avoidance of soda consumption and desserts). This diet also supports the acquisition of healthy eating habits characterized by higher consumption of fruits, vegetables, and whole grains, and encourages a reduction in the intake of saturated fat, sodium, added sugars, and canned foods. Limiting beverage consumption of water or fresh coconut water between meals is also encouraged. In this pilot study, the investigators hypothesized that the Gracie diet it could be an alternative option to improve GERD symptoms in those patients who do not respond to standard doses of PPI and/or H2 receptor antagonists.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at registration.
* Patients with ongoing symptoms of GERD: heartburn (pyrosis) mid-sternal chest pain, regurgitation of fluid or food, development of esophageal inflammation that may lead to swallowing dysfunction, or extraesophageal manifestations (i.e. cough, bronchospasms, and hoarseness).
* Use of one of the following PPI medications: omeprazole, lansoprazole, pantoprazole, rabeprazole, esomeprazole or dexlansoprazole. And/or use of one of the following H2 blockers medications as well: famotidine, cimetidine, ranitidine or nizatidine.
* Willing to comply with the Gracie diet regimen

Exclusion Criteria:

* Age < than 18 years.
* Patients unable to speak English.
* Pregnancy or nursing.
* Complicated oropharyngeal dysphagia or other condition with risk for aspiration from oral ingestion.
* Exclusion of other causes of symptoms as mechanical gastrointestinal obstruction, Barrett's esophagus and cancer of the esophagus by standard radiographic or endoscopic test evidenced in the medical record chart.
* A prior surgery of the upper gastrointestinal tract.
* Failure to give informed consent.
* Any other condition, which in the opinion of the investigator would impede compliance or hinder the completion of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in University of California Scleroderma Clinical Trial Consortium Gastrointestinal Tract (UCLA SCTC GIT 2.0) score | Baseline, week 2 and week 4
  The effect of the Gracie Diet in GERD symptoms by changes in the UCLA SCTC GIT 2.0 score.
  The UCLA-SCTC GIT 2.0 is a multi-item instrument that measures GI symptoms and the impact on health related quality of life. Includes 34 questions in 7 domains (reflux, distension, soilage, diarrhea, social function, emotional wellbeing and constipation) during a 7 day recall period. Each domain is weighted and scored, and a total score is then calculated.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) scale score | Baseline, week 2 and week 4
  The effect of the Gracie Diet in GERD symptoms by changes in the PROMIS Scale score. This questionnaire has items that measure the frequency, severity, impact, and bother of cardinal GERD symptoms, including heartburn and regurgitation, using a seven-day recall period. The questionnaire consists of 13 questions, and in each question, the answers are scored from 0 to 5.
Change in the Reflux Symptoms Index (RSI) score | Baseline, week 2 and week 4
  The effect of the Gracie Diet in GERD symptoms by changes in the RSI score. The RSI is a nine-item questionnaire assessing symptom severity, and designed to assess the severity of symptoms related to laryngopharyngeal reflux. Normative data suggests that a RSI of greater than or equal to 13 is clinically significant. Therefore a RSI > 13 may be indicative of significant reflux disease.
Change in the Health-related Quality Of Life scale for GERD (GERD-HRQL) score | Baseline, week 2 and week 4
  The effect of Gracie Diet in GERD symptoms by changes in the score of the GERD - HRQL. The GERD-HRQL was developed to survey symptomatic outcomes and therapeutic effects in patients with GERD. The scale has 11 items, which focus on heartburn symptoms, dysphagia, medication effects and the patient's present health condition. The GERD-HRQL takes approximately one minute to complete. Each item is scored from 0 to 5, with a higher score indicating a better QOL.
Change in the Gracie Diet adherence as assessed by a patient diary inventory | Daily up to 4 weeks
  Assess adherence to diet through the use of a diary where the patient can track the food eaten during the day.
Change in GERD medication | Baseline, week 2 and week 4
  The effect of Gracie Diet in medication intake through a review of the medication list, dose and intake frequency.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline, week 2 and week 4
  The effect of Gracie Diet in the BMI (kg/m^2). BMI is a person's weight in kilograms divided by the square of height in meters. The range values are Below 18.5 Underweight 18.5 - 24.9 Normal or Healthy Weight 25.0 - 29.9 Overweight 30.0 or higher Obese

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bulat, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No